CLINICAL TRIAL: NCT06115837
Title: Prognosis Stratification for pT4bN0M0 Colorectal Cancer Following Multivisceral Resection: A Multi-institutional Retrospective Analysis
Brief Title: Prognosis Stratification for pT4bN0M0 Colorectal Cancer Following Multivisceral Resection
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianqiang Tang, Associate professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC2330
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Multivisceral resection; Prognosis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: multivisceral resection — The prognostic factors were analyzed for pT4bN0M0 colorectal cancer after multivisceral resection

SUMMARY:
The purpose of this study was to identify the prognostic factors of affecting pT4bN0M0 colorectal cancer patients, so as to better stratify the prognostic differences among patients with the same stage.

DETAILED DESCRIPTION:
Patients with pT4b stage colorectal cancer (CRC) are a complex and special group due to the diversity of infiltrated organs, patients with the same stage often have different prognosis after multivisceral resection (MVR), some important prognostic factors have not been deeply explored, and additional prognostic factors are needed to improve the survival assessment of these patients. In this study, investigators attempted to evaluate the prognostic factors of pT4bN0M0 colorectal cancer, and then stratify the prognosis of such patients to distinguish the survival differences among different patients.

This study was a multicenter retrospective cohort study based on a multicenter database which contained hospitalization.The prognostic factors of pT4bN0M0 colorectal cancer patients were analyzed, and the prognostic grading system was constructed to accurately stratify the survival of pT4bN0M0 patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was pathologically diagnosed as colorectal adenocarcinoma.
2. Patients with pT4bN0M0 colorectal cancer.
3. Patients with R0 resection.

Exclusion Criteria:

1. Patients with distant metastasis.
2. Patients with R1 or R2 resection.
3. Patients with lymph node metastasis
4. Recurrent colorectal cancer.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient experienced multivisceral resection for pT4bN0M0 colorectal cancer from January 2010 to December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Overall survival | The endpoint of the overall survival assessment is the last follow-up or patient death. Follow-up time is up to 72 months.
  Overall survival is defined as the time from the surgery to death or last follow-up, regardless of disease recurrence, which was measured in months.
Cancer specific survival | The endpoint of the cancer specific survival assessment is the patient death due to cancer. Follow-up time is up to 72 months.
  Cancer specific survival is defined as the time from the diagnosis to death due to cancer progression, which was measured in months.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Quan J, Zuo K, Li G, Liu J, Mei S, Hu G, Qiu W, Zhuang M, Meng L, Wang X, Chang H, Tang J. Prognostic stratification of patients with pT4bN0M0 colorectal cancer following multivisceral resection: a multi-institutional case series analysis. Int J Surg. 2024 Sep 1;110(9):5323-5333. doi: 10.1097/JS9.0000000000001646. PMID 38768462